CLINICAL TRIAL: NCT05222126
Title: Efficacy of Ultrasound-Guided Hydrodissection in Patients With Carpal Tunnel Syndrome
Brief Title: Efficacy of Ultrasound-Guided Hydrodissection in Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Nuran Eyvaz, Asistant Profesor, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTSHD22
Record Dates: First submitted 2022-01-31; First posted 2022-02-03 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Musculoskeletal Diseases; Median Nerve Disease; Carpal Tunnel Syndrome; Ultrasound-Guided Injection
Keywords: Carpal Tunnel Syndrome; Ultrasound-Guided Injection; Hydrodissection
MeSH Terms: conditions — Musculoskeletal Diseases; Median Neuropathy; Carpal Tunnel Syndrome | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ultrasound-guided Hydrodissection (HD) with 5 cc 5% Dextrose (Experimental): The median nerve will be defined at the proximal entrance of the carpal tunnel (scaphoid-pisiform plane). Under the ulnar approach with the in-plane technique, it was planned to hydrodissect the median nerve using 5 cc of 5% dextrose.
  Interventions: Procedure: Ultrasound-guided Hydrodissection (HD) with 5 cc 5% Dextrose
- Ultrasound-guided Hydrodissection (HD) with 5 cc Normal Saline (Active Comparator): The median nerve will be defined at the proximal entrance of the carpal tunnel (scaphoid-pisiform plane). Under the ulnar approach with the in-plane technique, it was planned to hydrodissect the median nerve , using 5 cc normal saline.
  Interventions: Procedure: Ultrasound-guided Hydrodissection (HD) with 5 cc Normal Saline
- Ultrasound-guided Hydrodissection (HD) with 10 cc 5% Dextrose (Experimental): The median nerve will be defined at the proximal entrance of the carpal tunnel (scaphoid-pisiform plane). Under the ulnar approach with the in-plane technique, it was planned to hydrodissect the median nerve , using 10 cc 5% dextrose.
  Interventions: Procedure: Ultrasound-guided Hydrodissection (HD) with 10 cc 5% Dextrose
- Ultrasound-guided Hydrodissection (HD) with 10 cc Normal Saline (Active Comparator): The median nerve will be defined at the proximal entrance of the carpal tunnel (scaphoid-pisiform plane). Under the ulnar approach with the in-plane technique, it was planned to hydrodissect the median nerve from , using 10 cc normal saline.
  Interventions: Procedure: Ultrasound-guided Hydrodissection (HD) with 10 cc Normal Saline

INTERVENTIONS:
Procedure: Ultrasound-guided Hydrodissection (HD) with 5 cc 5% Dextrose — The median nerve will be defined at the proximal entrance of the carpal tunnel (scaphoid-pisiform plane). Under the ulnar approach with the in-plane technique, first it was planned to hydrodissect the median nerve from the retinaculum superiorly and then from the flexor tendons inferiorly, using 5 cc of 5% dextrose.
  Arms: Ultrasound-guided Hydrodissection (HD) with 5 cc 5% Dextrose
Procedure: Ultrasound-guided Hydrodissection (HD) with 5 cc Normal Saline — The median nerve will be defined at the proximal entrance of the carpal tunnel (scaphoid-pisiform plane). Under the ulnar approach with the in-plane technique, first it was planned to hydrodissect the median nerve from the retinaculum superiorly and then from the flexor tendons inferiorly, using 5 cc normal saline.
  Arms: Ultrasound-guided Hydrodissection (HD) with 5 cc Normal Saline
Procedure: Ultrasound-guided Hydrodissection (HD) with 10 cc 5% Dextrose — The median nerve will be defined at the proximal entrance of the carpal tunnel (scaphoid-pisiform plane). Under the ulnar approach with the in-plane technique, first it was planned to hydrodissect the median nerve from the retinaculum superiorly and then from the flexor tendons inferiorly, using 10 cc 5% dextrose.
  Arms: Ultrasound-guided Hydrodissection (HD) with 10 cc 5% Dextrose
Procedure: Ultrasound-guided Hydrodissection (HD) with 10 cc Normal Saline — The median nerve will be defined at the proximal entrance of the carpal tunnel (scaphoid-pisiform plane). Under the ulnar approach with the in-plane technique, first it was planned to hydrodissect the median nerve from the retinaculum superiorly and then from the flexor tendons inferiorly, using 10 cc normal saline.
  Arms: Ultrasound-guided Hydrodissection (HD) with 10 cc Normal Saline

SUMMARY:
The aim of our study is to determine the effectiveness of US-guided hydrodissection of the median nerve in different contents and volumes in patients diagnosed with mild to moderate carpal tunnel syndrome.

DETAILED DESCRIPTION:
Carpal tunnel syndrome is the most common form of entrapment neuropathies. Anatomically, the roof of the carpal tunnel consists of carpal bones, it is located under the transverse carpal ligament, and there are 9 tendon packs of the forearm flexors and the median nerve. Clinically, sensory (paresthesia and hypoesthesia), motor deficits and pain occur in the distribution of the median nerve secondary to mechanical compression and local ischemia.

Conservative treatment options are available for patients diagnosed with mild and moderate CTS as a result of CTS classification. Treatment options for symptom relief include physical therapy applications, splinting, and wrist injections. Among local injection treatments; applications such as corticosteroids and local anesthetics are included.

Ultrasound-guided injections of peripheral nerves are generally superior to blind injections as they prevent damage to critical vascular structures in the surrounding tissue accompanying the nerves and reduce the risk of intraneural injections.

Ultrasound (US) guided hydrodissection of peripheral nerves (HD) is a technique that uses high-resolution ultrasound-guided fluid injection to separate nerves from a surrounding or adjacent structure, usually fascia. The aim is to restore function to the nerve and to release soft tissue adhesions that cause entrapment.

This investigation was designed double-blind prospective randomized study. Participants were randomized into 4 groups: Ultrasound-guided Hydrodissection (HD) with 5 cc 5% dextrose, Ultrasound-guided Hydrodissection (HD) with 5 cc normal saline, Ultrasound-guided Hydrodissection (HD) with 10 cc 5% dextrose, Ultrasound-guided Hydrodissection (HD) with 10 cc normal saline.

Ultrasonographic evaluation and ultrasound-guided injection were planned to be performed with the 10-18-MHz linear probe of the MyLab 70 (Esaote, Genova, Italy) device by a physician experienced in US. It was designed in such a way that the physician was blind to the clinical information of the patients and the injected material.

As evaluation parameters, Visual Analogue Scale (VAS), Boston Carpal Tunnel Syndrome Questionnaire (BCTQ), Cross-sectional Area of Median Nerve (CSA), Hand and finger grip strength assessment, and Electrophysiological assessment will be evaluated. It was planned that the evaluations were made and recorded by a blinded physician to the groups at the beginning of the treatment, at the 1st month and at the 3rd month controls.

ELIGIBILITY:
Inclusion Criteria:

* Presence of symptoms of carpal tunnel syndrome, including nocturnal, postural, or movement-related paresthesias +/- pain in the median nerve distribution area in the hand for more than 3 months
* Presence of mild to moderate carpal tunnel syndrome proven by electrophysiological study
* Loss of sensation with numbness in the median nerve-innervated areas of the hand, weakness of the median nerve-innervated thenar muscles
* Positive Phalen test and/or Tinel sign

Exclusion Criteria:

* Patients who can mimic the diagnosis of carpal tunnel syndrome, such as cervical radiculopathy, polyneuropathy, brachial plexopathy, thoracic outlet syndrome
* Patients who have had an injection into the carpal tunnel in the last 6 months
* Patients with thenar muscle atrophy
* History of Carpal tunnel surgery
* Regular use of systemic nonsteroidal anti-inflammatory drugs and corticosteroids
* Pregnancy
* Rheumatoid arthritis, systemic lupus erythematosus, gout, systemic sclerosis, dermatomyositis, polymyositis
* Presence of malignancy
* Presence of active infection

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | up to 12th week
  Pain intensity was measured with visual analogue scale for pain (0-10 mm; 0 means no pain, 10 means severe pain) which is used to measure musculoskeletal pain with very good reliability and validity.

SECONDARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) | up to 12th week
  The Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) is a frequently used questionnaire for CTS that includes 2 components. It evaluates for grading under two sub-headings: symptom severity scale (11 questions) and functional status scale (8 questions). Scores range from 0 to 5 for each question; 0 represents no difficulty during the activity, 5 represents extremely severe dysfunction.
Cross-sectional area of the Median Nerve (CSA) | up to 12th week
  The cross-sectional area (CSA) of the median nerve will be used for analysis by the mean value of 3 measurements made with an electronic caliper at the same level as the injection site (scaphoid-pisiform level).
  CSA values increase as clinical findings worsen.
Electrophysiological Evaluation | up to 12th week
  Antidromic sensory nerve conduction velocity and distal motor latency of the median nerve will be measured in all patients. All measurements will be made 3 times and the average value will be taken. To diagnose CTS electrophysiologically; The median nerve peak sensory conduction velocity recorded antidromically from the second finger should be slower than 41.25 m/sec, the conduction velocity should be slower than 34 m/sec in the mixed nerve conduction study in the palm-wrist segment (8 cm), and/or recordings from the APB (abductor pollicis brevis) muscle DML (distal motor latency) was determined to be longer than 3.8 ms with stimulation of the median nerve from the wrist segment (5 cm).
Hand and Finger Grip Strength Assessment | up to 12th week
  The hand grip strength of the participants will be measured with the "Jamar Hand Dynamometer". Measurements will be made with the shoulder in adduction and neutral rotation adjacent to the trunk, elbow 90 degrees flexed, wrist 0-30 degrees dorsiflexion and 0-15 degrees ulnar deviation with thumb up. Finger grip strength will be evaluated with the "Jamar Digital Pinchmeter". Patients will be placed in the sitting position with the wrist in 90° flexion and the forearm in the neutral position. Measurements will be made bilaterally in three different positions as lateral, palmar and fingertip grips. Patients will be asked to squeeze with maximum force and each measurement will be made three times, and their averages will be recorded in kg. The dynamometer has a dual scale readout which displays isometric grip force from 0-90 kg. Higher scores means better grip strength.

CONTACTS AND LOCATIONS:
Overall Officials: Nuran EYVAZ, MD, Principal Investigator — Afyonkarahisar Health Sciences University; Ali İzzet AKÇİN, MD, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Afyonkarahisar Health Sciences University, Afyonkarahisar, Afyonkarahi̇sar, Turkey (Türkiye)

REFERENCES:
- [Background] Babaei-Ghazani A, Forogh B, Raissi GR, Ahadi T, Eftekharsadat B, Yousefi N, Rahimi-Dehgolan S, Moradi K. Ultrasound-Guided Corticosteroid Injection in Carpal Tunnel Syndrome: Comparison Between Radial and Ulnar Approaches. J Pain Res. 2020 Jun 26;13:1569-1578. doi: 10.2147/JPR.S248600. eCollection 2020. PMID 32617017
- [Background] Chang KV, Wu WT, Ozcakar L. Ultrasound imaging and guidance in peripheral nerve entrapment: hydrodissection highlighted. Pain Manag. 2020 Mar;10(2):97-106. doi: 10.2217/pmt-2019-0056. Epub 2020 Mar 12. PMID 32162601
- [Background] Lam KHS, Hung CY, Chiang YP, Onishi K, Su DCJ, Clark TB, Reeves KD. Ultrasound-Guided Nerve Hydrodissection for Pain Management: Rationale, Methods, Current Literature, and Theoretical Mechanisms. J Pain Res. 2020 Aug 4;13:1957-1968. doi: 10.2147/JPR.S247208. eCollection 2020. PMID 32801851
- [Derived] Eyvaz N, Adar S, Akcin AI, Dundar U, Toktas H, Eroglu S. Comparison of Ultrasound-Guided Hydrodissection With Various Volumes of 5% Dextrose for Carpal Tunnel Syndrome: A Prospective Randomized Controlled Double-Blind Trial. Am J Phys Med Rehabil. 2025 Jul 1;104(7):596-604. doi: 10.1097/PHM.0000000000002675. Epub 2024 Dec 3. PMID 39642354